CLINICAL TRIAL: NCT03504670
Title: Preterm Induction of Labor Timing of Amniotomy: A Randomized Controlled Trial
Acronym: PITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lindsay Speros Robbins, MD, MPH, Instructor-Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB_EarlyAROM
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Preterm Pregnancy; Labor Induction
Keywords: Labor induction; Cesarean delivery; Preterm labor induction; Duration of labor induction

STUDY DESIGN:
Intervention Model Description: Participants are assigned to early amniotomy (<4cm cervical dilation) or late amniotomy (≥4cm dilated). Participants may crossover due due to clinical conditions that are not preventable. These conditions may include: unengaged vertex at time of attempted amniotomy, need for internal monitors, or cervical dilation that does not reach 4cm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early amniotomy (Experimental): Women randomized to early amniotomy will have their membranes ruptured in usual fashion using an amniotomy hook when the cervix is less than 4cm dilated. This will occur after cervical ripening has taken place, with 1) a cervical Foley balloon catheter with or without oxytocin and/or 2) misoprostol. Prior to amniotomy, the obstetric provider will assess whether or not the fetal head is engaged. If the fetal head is not engaged (applied to the cervix), amniotomy will be deferred. The patient will be examined every 2 hours until amniotomy can be safely performed (in keeping with our institutional standard of care to examine women every 2-4 hours in labor).
  Interventions: Procedure: Early Amniotomy
- Late amniotomy (Experimental): Women randomized to late amniotomy will have their membranes ruptured once the cervix reaches at least 4cm dilation. This will occur after cervical ripening has taken place, with 1) a cervical Foley balloon catheter with or without oxytocin and/or 2) misoprostol. If the cervix fails to reach 4cm dilation 12 hours following cervical ripening, amniotomy will be performed.
  Interventions: Procedure: Late Amniotomy

INTERVENTIONS:
Procedure: Early Amniotomy — This intervention involves using an amniotomy hook to rupture the membranes during a sterile vaginal exam. This intervention will be performed prior to the cervix being dilated 4cm.
  Arms: Early amniotomy
Procedure: Late Amniotomy — This intervention involves using an amniotomy hook to rupture the membranes during a sterile vaginal exam. This intervention will be performed once the cervix is at least 4cm dilated.
  Arms: Late amniotomy

SUMMARY:
Artificial rupture of membranes (amniotomy) is a commonly used technique to safely induce and augment labor. It has been shown to reduce the duration of spontaneous and induced labor in term patients (≥37 weeks' gestation). The utility of amniotomy in preterm patients (<37 weeks' gestation) undergoing medically-indicated induction of labor is unknown. However, it remains a commonly used strategy. We will conduct a trial comparing early amniotomy versus late amniotomy during medically-indicated induction of labor between 23.0 and 35.6 weeks gestation. Women will be randomized to early or late amniotomy after the obstetrician has decided to induce labor for a medical indication. We hypothesize that more women in the early amniotomy group will require cesarean delivery, and the duration of labor will increase in the early amniotomy group.

DETAILED DESCRIPTION:
The rate of preterm birth in the United States is nearly 10%. Up to one-third of these births are the result of a medically-indicated delivery. While induction of labor in women at term gestation has been extensively studied, the same is not true for preterm gestations. Consequently, the same methods of labor induction are used in term and preterm gestations, although preterm gestations may have different responses to induction agents compared to term gestations.

At our institution, a standard induction of labor - for term or preterm women - is performed using a cervical Foley catheter or misoprostol for cervical ripening with the addition of intravenous oxytocin for labor augmentation. As membranes do not typically spontaneously rupture during the induction process, amniotomy is commonly utilized by providers to help augment labor. Amniotomy releases prostaglandin-rich amniotic fluid. These prostaglandins are important mediators of uterine contractility and ultimately active labor. It has been shown to reduce the duration of spontaneous and induced labor in term patients.

The timing of amniotomy is left up to the discretion of the treating providers, as there are no randomized controlled trials to support early versus late amniotomy at preterm gestations. However, a retrospective cohort of nulliparous and multiparous women at our institution undergoing induction at 23-34 weeks, and evaluating early amniotomy at <4cm cervical dilation versus late amniotomy at ≥4cm dilation, showed an increased risk of cesarean delivery and increased time from start of induction to delivery for early amniotomy, although only the cesarean delivery outcome was significant after adjusting for confounders.

We will conduct an intention-to-treat randomized controlled trial comparing early amniotomy versus late amniotomy during medically-indicated induction of labor between 23.0 and 35.6 weeks gestation. Women will be randomized to early or late amniotomy after the attending obstetrician has decided to induce labor for a medical indication. Early amniotomy will be performed prior to 4cm cervical dilation being reached. Late amniotomy will be performed at greater than or equal to 4cm cervical dilation.

The purpose of this study is to determine whether timing of amniotomy during medically-indicated preterm induction of labor affects labor outcomes. We will specifically be looking at risk of cesarean delivery, duration of labor, maternal morbidity, and neonatal morbidity. We hypothesize that more women in the early amniotomy group will require cesarean delivery and that the duration of labor will increase in the early amniotomy group.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Gestational age at randomization between 23.0 and 35.6 weeks
* Induction of labor planned for maternal or fetal indications
* Reassuring fetal status
* Vertex presentation

Exclusion Criteria:

* Plan for cesarean delivery or contraindication to labor
* Cervix ≥4cm dilated at start of induction
* Signs of spontaneous labor (active contractions with cervical change)
* Ruptured membranes
* Chorioamnionitis
* Intrauterine fetal demise
* Known major fetal anomaly
* Participation in any other clinical trial involving the course of labor
* Maternal hepatitis B, C, or HIV infection (or unknown status)
* Deferring intrapartum fetal monitoring and/or cesarean section for any reason (for example, after periviability counseling)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Cesarean delivery | Duration is dependent upon the length of labor. The maximum time frame would be anticipated to be 120 hours from start of the induction.
  Proportion of women requiring cesarean delivery

SECONDARY OUTCOMES:
Interval from induction onset to delivery | Duration is dependent upon the length of labor. The maximum time frame would be anticipated to be 120 hours from start of the induction.
  Time (hours) from the start of induction (initiation of first cervical ripening agent) to delivery (vaginal or cesarean)
Interval from induction onset to vaginal delivery | Duration is dependent upon the length of labor. The maximum time frame would be anticipated to be 120 hours from start of the induction.
  Time (hours) from the start of induction (initiation of first cervical ripening agent) to vaginal delivery only
Composite maternal morbidity | Measured from start of induction of labor up to 42 days following delivery
  Composed of seven outcomes:
  1. chorioamnionitis (defined as maternal fever >100.3 plus maternal tachycardia, fetal tachycardia, purulent amniotic fluid, or fundal tenderness prior to delivery)
  2. endometritis (defined as maternal fever >100.3 at least 12 hours after delivery with fundal tenderness or purulent discharge)
  3. surgical site infection (infection within 30 days at the surgical site including superficial, deep, organ/space infections)
  4. pneumonia (radiologic diagnosis of pneumonia accompanied by clinical signs/symptoms)
  5. urinary tract infection (>100,000 colonies of a single species in urine culture accompanied by clinical signs/symptoms)
  6. postpartum hemorrhage (estimated blood loss >1000 mL)
  7. umbilical cord prolapse
Composite neonatal morbidity | Measured up to 28 days of life for the newborn
  Composed of five outcomes:
  1. perinatal death (death of a fetus during labor or within 28 days of life)
  2. neonatal sepsis (critically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal X-ray confirming infection)
  3. intraventricular hemorrhage (confirmed on ultrasound or MRI)
  4. cord blood acidemia (umbilical artery gas pH <= 7.0 or base excess >= 12)
  5. Apgar <5 at 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay S Robbins, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmigham, Women and Infants' Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Fraser WD, Marcoux S, Moutquin JM, Christen A. Effect of early amniotomy on the risk of dystocia in nulliparous women. The Canadian Early Amniotomy Study Group. N Engl J Med. 1993 Apr 22;328(16):1145-9. doi: 10.1056/NEJM199304223281602. PMID 8257472
- [Background] Gagnon-Gervais K, Bujold E, Iglesias MH, Duperron L, Masse A, Mayrand MH, Sansregret A, Fraser W, Audibert F. Early versus late amniotomy for labour induction: a randomized controlled trial. J Matern Fetal Neonatal Med. 2012 Nov;25(11):2326-9. doi: 10.3109/14767058.2012.695819. Epub 2012 Jun 13. PMID 22616980
- [Background] Macones GA, Cahill A, Stamilio DM, Odibo AO. The efficacy of early amniotomy in nulliparous labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):403.e1-5. doi: 10.1016/j.ajog.2012.08.032. Epub 2012 Aug 24. PMID 22959833
- [Background] Onah LN, Dim CC, Nwagha UI, Ozumba BC. Effect of early amniotomy on the outcome of spontaneous labour: a randomized controlled trial of pregnant women in Enugu, South-east Nigeria. Afr Health Sci. 2015 Dec;15(4):1097-103. doi: 10.4314/ahs.v15i4.7. PMID 26958009
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Parrish MM, Kuper SG, Jauk VC, Baalbaki SH, Tita AT, Harper LM. Does Early Artificial Rupture of Membranes Speed Labor in Preterm Inductions? Am J Perinatol. 2018 Jul;35(8):716-720. doi: 10.1055/s-0037-1612631. Epub 2017 Dec 14. PMID 29241279
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Kuper SG, Sievert RA, Steele R, Biggio JR, Tita AT, Harper LM. Maternal and Neonatal Outcomes in Indicated Preterm Births Based on the Intended Mode of Delivery. Obstet Gynecol. 2017 Nov;130(5):1143-1151. doi: 10.1097/AOG.0000000000002320. PMID 29016494
- [Background] Cooney LG, Bastek JA. The Association between Early Artificial Amniotomy and Chorioamnionitis in Nulliparous Induction of Labor. Int Sch Res Notices. 2014 Dec 16;2014:628452. doi: 10.1155/2014/628452. eCollection 2014. PMID 27379338